CLINICAL TRIAL: NCT01244100
Title: Food-Effect Pharmacokinetic Study of PL2200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Jason Moore, Vice President, PLx Pharma Inc.
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: PL-ASA-003
Record Dates: First submitted 2010-10-25; First posted 2010-11-19 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Food-effects PK study in healthy subjects.

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- PL2200 (Experimental)
  Interventions: Drug: PL2200 fasted; Drug: PL2200 fed

INTERVENTIONS:
Drug: PL2200 fasted — Fasted state
Drug: PL2200 fed — Fed state

SUMMARY:
This trial is a food-effect study to assess fasted versus fed pharmacokinetics of PL2200.

ELIGIBILITY:
Inclusion Criteria:

* Healthy normal male and female volunteers between 21 and 65 years of age.

Exclusion Criteria:

* Abnormal findings on physical examination or clinical laboratories, or significant medical history.
* Subject with hypersensitivity or contraindications to aspirin, ibuprofen, or other nonsteroidal anti-inflammatory drug (NSAID).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Effect of food by ratio of least-squares means (LSM) of the pharmacokinetic (PK) parameter of AUC0-t of the primary metabolite, salicylic acid, in the fed state versus the fasted state. | 24 hours
Effect of food by ratio of least-squares means (LSM) of the PK parameter of AUC0-inf of the primary metabolite, salicylic acid, in the fed state versus the fasted state. | 24 hours
Effect of food by ratio of least-squares means (LSM) of the PK parameter of Cmax of the primary metabolite, salicylic acid, in the fed state versus the fasted state. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Upendra K Marathi, PhD, Study Director — PLx Pharma Inc.
Locations (1):
- Houston Institute for Clinical Research, Houston, Texas, United States

REFERENCES:
- [Derived] Angiolillo DJ, Bhatt DL, Lanza F, Deliargyris EN, Prats J, Fan W, Marathi U. Bioavailability of aspirin in fasted and fed states of a novel pharmaceutical lipid aspirin complex formulation. J Thromb Thrombolysis. 2020 Apr;49(3):337-343. doi: 10.1007/s11239-020-02051-5. PMID 32080811